CLINICAL TRIAL: NCT07402473
Title: EUREKA Study: Phase 2 Study to Optimize Neoadjuvant Therapy in HER2-positive Early-stage Breast Cancer Using ctDNA and HARPS Biomarker Assay
Brief Title: EUREKA Study:Phase 2 Study to Optimize Neoadjuvant Therapy in HER2-positive Early-stage Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Mridula George, MD, Associate Program Director, Breast, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 042507; Pro2025002581 (Other: Rutgers Institutional Review Board)
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: HER2-positive Early-stage Breast Cancer
MeSH Terms: interventions — Trastuzumab; pertuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: The study is a single arm phase 2 study, which will evaluate optimization of neoadjuvant chemotherapy in patients with stage II-III HER2-positive breast cancer. Tumors will undergo testing using HARPS assay to identify HARPS-positive HER2-positive breast cancers. Patients will also have ctDNA monitored to identify patients that are at increased risk of recurrence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HARPS POSITIVE COHORT (Experimental): Arm A HARPS POSITIVE COHORT
  PART A:
  Patients with HARPS positive HER2 positive breast cancer will be treated with trastuzumab and pertuzumab for three cycles.
  PART B:
  Patients who have adequate treatment response after 3 cycles, continue trastuzumab and pertuzumab every 3 weeks for a minimum of 8 cycles in the neoadjuvant setting
  ARM B:
  HARPS-NEGATIVE COHORT
  Patients with HARPS negative tumors must have baseline detectable ctDNA. If patients do not have detectable ctDNA, they will be taken off study. These patients will be replaced.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Docetaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab is a targeted antibody therapy used to treat HER2-positive breast and stomach cancers by blocking the growth-stimulating HER2 protein
Drug: Pertuzumab — targeted therapy, a monoclonal antibody, used with other drugs (like trastuzumab and chemotherapy) to treat HER2-positive breast cancer, blocking HER2 proteins on cancer cells to stop their growth, and used for metastatic, locally advanced, or early-stage high-risk cases before or after surgery
Drug: Docetaxel — will be used with HARPS Negative: intravenous chemotherapy medication used to treat breast, lung, prostate, gastric, and head/neck cancers
Drug: Carboplatin — will be used with HARPS Negative: a platinum-based chemotherapy drug used primarily to treat advanced ovarian cancer, often in combination with other agents, as well as lung, head and neck, and brain cancers

SUMMARY:
This is an open-label phase 2 study to evaluate the pCR rate in patients diagnosed with HER2 positive breast cancer treated on an adaptive clinical trial design.

Tumors will undergo testing using a novel molecular phosphoprotein-based biomarker assay, HER2 Activation Response Predictive Signature (HARPS) to identify HARPS-positive breast cancers.

To assess 3-year invasive disease-free survival (iDFS) in patients with HARPS-positive and HARPS-negative HER2-positive breast cancer.

To correlate changes in ctDNA with treatment outcomes in patients with HARPS-positive and HARPS-negative HER2-positive breast cancer.

To understand the changes in quality of life (QOL) measure in patients with HARPS-positive HER2-positive breast cancer treated using an adaptive neoadjuvant trial design.

DETAILED DESCRIPTION:
EUREKA is a phase II study that will evaluate optimization of neoadjuvant therapy in patients with stage II-III HER2-positive breast cancer. This adaptive clinical trial will enroll patients with cT2-T3 N0-2 HER2-positive breast cancer. Tumors will undergo testing using HARPS assay to identify HARPS-positive and HARPS negative HER2-positive breast cancers.

Patients with HARPS-positive HER2-positive breast cancer will be treated using an adaptive trial design to optimize neoadjuvant therapy such we are maximizing treatment efficacy while reducing risk of treatment related toxicities. Patient will be treated with dual HER2-targeted therapy (trastuzumab and pertuzumab) for 3 cycles. Treatment response will be monitored by ctDNA and MRI breast. If there is treatment response, patients will be treated with 6 cycles of trastuzumab and pertuzumab. If there is no treatment response after 6 weeks, then patients will be treated with the addition of single agent chemotherapy (docetaxel/paclitaxel/Abraxane) with trastuzumab/pertuzumab for 4 cycles followed by 2 cycles of trastuzumab and pertuzumab. Then patients will proceed with breast surgery.

Patients with HARPS-negative HER2-positive breast cancer and detectable ctDNA at time of diagnosis will be treated with 4 cycles of Taxane, platinum, trastuzumab and pertuzumab, and they will be monitored with ctDNA for ctDNA clearance. Patients who have ctDNA clearance will be treated with additional 2 cycles of the same regimen and then proceed to have surgery. If patients have detectable ctDNA at 12 weeks, then neoadjuvant therapy will be escalated to add anthracycline based regimen or trastuzumab deruxtecan (T-DXD) pe treating physicians choice.

The study will enroll a total of 50 patients- 25 patients with HARPS-positive HER2-positive early-stage breast cancer and 25 patients with HARPS-negative HARPS-positive early-stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Tumor size greater than 2cm or lymph node positive by imaging or clinical exam (cT2-T3 N0-2)
  2. Tumors must be HER2 positive either by IHC (3+) or by IHC 2+ and FISH positive.
  3. Patient must have known estrogen receptor (ER) and progesterone receptor (PR) status locally determined prior to study entry
  4. Patient must have adequate tumor for HARPS testing.
  5. Patients must have ctDNA collection prior to treatment on trial.
  6. Patient must be able to do breast MRI as determined by the study
  7. Baseline LVEF > 50% (Most recent within the last 5 years)
  8. No prior history of systemic treatment with anthracyclines-based chemotherapy.
  9. Adequate bone marrow function:

     * ANC ≥ 1500/uL
     * platelet count ≥ 100,000/uL
     * hemoglobin ≥ 9.0 g/dL
  10. Adequate hepatic function:

      * Total bilirubin ≤ 1.5 X ULN
      * AST (SGOT) ≤ 5 X ULN
      * ALT (SGPT) ≤ 5 X ULN
  11. Patients with biliary obstruction must have restored biliary flow by placement of an endoscopic common bile duct stent or a percutaneous drainage.
  12. Adequate renal function, Creatinine < 1.5x institutional ULN or calculated creatinine clearance ≥ 50 mL/min as estimated using the Cockcroft-Gault formula.
  13. Ability to understand the nature of this study protocol and give written informed consent.
  14. Willingness and ability to comply with scheduled visits and treatment plans
  15. Prior cancers allowed if no evidence of disease in last 5 years. Prior history of ipsilateral invasive breast cancers are not allowed.

Exclusion Criteria:

1. Previous treatment with chemotherapy, anti-HER2 therapy, radiation therapy, or endocrine therapy for invasive breast cancer. Exception: patients can start upto 1 cycle of HP prior to starting treatment on study.
2. cT4 and/or cN3 tumors
3. Evidence of metastatic disease by routine clinical assessment
4. Bilateral breast cancer
5. History of other malignancy within the last five years prior to first dose of study drug administration, except for curatively treated basal and squamous cell carcinoma of the skin and/or in situ cervical carcinoma
6. Left ventricular ejection fraction (LVEF) below 50% as determined by multiple-gated acquisition (MUGA) scan or echocardiography (ECHO)
7. No active liver disease.
8. Any condition including the presence of laboratory abnormalities, which, in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study.
9. Pre-existing sensory neuropathy > grade 1.
10. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
11. Serious non-healing wound, ulcer, or bone fracture
12. Patient with uncontrolled and/ or active infection with HIV, Hepatitis B or Hepatitis C.
13. Patient who has a history of allergy or hypersensitivity to any of the study drugs.
14. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
outcomes that correspond directly to the objective(s) | up to 36 months
  The HARPS assay will be used to identify patients with HARPS positive and HARPS-negative HER2-positive breast cancer. Patients with Stage I-III who meet the specified eligibility criteria would be enrolled in the adaptive clinical trial.
  The study aims to understand whether the HARPS assay can help optimize the treatment regimen for patients diagnosed with HER2 positive breast cancer.
  The study will evaluate the pCR rates in patients treated with the adaptive trial regimen. The hypothesis of the study is that the adaptive treatment regimen will help improve pCR rates in patients diagnosed HER2-positive breast cancer based on the HARPS status of the tumor.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - RWJBarnabas Health - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - RWJBarnabas Health - Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Somerset, Somerville, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey